CLINICAL TRIAL: NCT05234684
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter Study Evaluating the Efficacy and Safety of Orelabrutinib Plus R-CHOP Versus Placebo Plus R-CHOP in Treatment-naïve Patients With MCD Subtype DLBCL
Brief Title: A Study of Orelabrutinib Plus R-CHOP in Treatment-naïve Patients With MCD Subtype Diffuse Large B-cell Lymphoma
Acronym: BELIEVE-01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICP-CL-00115
Record Dates: First submitted 2022-01-29; First posted 2022-02-10 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — orelabrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orelabrutinib+ R-CHOP (Experimental): Participants will receive 150 mg of oral orelabrutinib once daily with R-CHOP on day 1 of each cycle (21 days).
  Interventions: Drug: Orelabrutinib + R-CHOP
- Placebo+ R-CHOP (Placebo Comparator): Participants will receive 150 mg placebo once daily with R-CHOP on day 1 of each cycle (21 days).
  Interventions: Drug: Placebo + R-CHOP

INTERVENTIONS:
Drug: Orelabrutinib + R-CHOP — The orelabrutinib is a white, round, uncoated tablet. The R-CHOP include rituximab, cyclophosphamide, doxorubicin, vincristine, and prednison.
  Other Names: ICP-022+ R-CHOP
  Arms: Orelabrutinib+ R-CHOP
Drug: Placebo + R-CHOP — The placebo is a white, round, uncoated tablet. The R-CHOP include rituximab, cyclophosphamide, doxorubicin, vincristine, and prednison.
  Arms: Placebo+ R-CHOP

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of orelabrutinib combined with R-CHOP regimen versus placebo with R-CHOP in the treatment of treatment-naïve patients with MCD subtype DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 18 and 80 years old
2. Treatment-naive patients
3. Histologically confirmed diffuse large B-cell lymphoma (DLBCL) and CD20 positive.
4. Provide FFPE slices of past or fresh tumor biopsy tissue.
5. At least one measurable lesion.
6. Lymphoma International Prognostic Score (IPI) ≥ 2.
7. Ann Arbor stage II-IV, or stage I with bulky lesion (diameter > 7.5 cm）
8. ECOG PS score of 0-2
9. Subjects who in line with the testing standard of the clinical trial laboratory.
10. Life expectancy ≥ 6 months.
11. Able to provide signed written informed consent.

Exclusion Criteria:

1. History of other active malignancies within 5 years of study entry, unless cured without evidence of relapse or metastasis
2. Lymphoma involving the central nervous system or leptomeningeal metastasis.
3. Transformed lymphoma, that is transformed from other types of lymphoma.
4. Primary mediastinal large B-cell lymphoma.
5. History of stroke or intracranial hemorrhage within 6 months before screening.
6. Co-morbidity of uncontrolled or significant cardiovascular disease, significant impaired lung function, significant gastrointestinal abnormalities, uncontrolled infections (including HBV, HCV, HIV/AIDS and tuberculosis), or active autoimmune disease.
7. Active bleeding within 2 months before screening, or a clear bleeding tendency determined by the investigator; a history of deep vein thrombosis or pulmonary embolism.
8. Previous history of surgeries (major 4 weeks and minor 2 weeks prior screening) , organ transplant or hematopoietic stem cell transplantation, or progressive multifocal leukoencephalopathy (PML).
9. Administer live and attenuated vaccines (semi-inactivated) within 28 days prior to first receiving the test drug.
10. Planned stem cell transplant during the experimental treatment are excluded.
11. Chemotherapy, immunotherapy, targeted therapy, radiotherapy, or traditional Chinese medicine with anti-tumor effects for the purpose of anti-tumor therapy within 4 weeks before starting to take the experimental drug. Excluding short-term emergency use of corticosteroids before treatment.
12. Current diagnosis of any mental or cognitive impairment, drug abuse, or alcohol abuse.
13. Pregnant, lactating women, or women at childbearing ages who will not use contraception during the study up to 12 months after the last dose of rituximab or 180 days after the last dose of study drug
14. The last use of strong CYP3A inhibitor or strong CYP3A inducer is less than 5 halflivesfrom the first trial drug, or the drug or food with moderate and strong CYP3A inhibitory effect or strong CYP3A induction effect is planned to be taken at the same time during this study.
15. Any serious medical condition that, in the investigator's opinion, would put the subject at unacceptable risk and/or would prevent the subject from signing the informed consent form. In the opinion of the investigator, the subject's participation in the study would be at unacceptable risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 3 years and 9 months
  Progression free survival (PFS) accessed by independent review committee (IRC)
Complete response rate (CRR) by independent review committee (IRC) | Up to 3 years and 9 months
  Complete response rate (CRR) at the completion of combination therapy accessed by independent review committee (IRC)

SECONDARY OUTCOMES:
Complete response rate (CRR) by investigator | Up to 3 years and 9 months
  Complete response rate (CRR) at the completion of combination therapy accessed by investigator
Overall response rate (ORR) by independent review committee (IRC) and investigator | Up to 3 years and 9 months
  Overall response rate (ORR) accessed by independent review committee (IRC) and investigator
Overall response rate (ORR) at the completion of combination therapy by independent review committee (IRC) and investigator | Up to 3 years and 9 months
  Overall response rate (ORR) at the completion of combination therapy accessed by independent review committee (IRC) and investigator
Duration of Response (DOR) | Up to 3 years and 9 months
  Duration of Response (DOR) accessed by independent review committee (IRC) and investigator
Disease free survival (DFS) rate and event free survival (EFS) rate | Up to 2 years
  2-year disease free survival (DFS) rate and 2-year event free survival (EFS) rate
Overall survival (OS) rate | Up to 2 years
  2-year overall survival (OS) rate Accessed by independent review committee (IRC) and investigator
Occurrence of adverse events and serious adverse events according to CTCAE V5.0. | Up to 3 years and 9 months
  The safety of Orelabrutinib measured by the occurrence of adverse events and serious adverse events according to CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Principal Investigator — Ruijin Hospital
Locations (44):
- China (44):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Anhui Provincal Cancer Hospital, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The Southwest Hospital of AMU, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital Of XIAMEN University, Xiamen, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - PEKING University SHENZHEN Hospital, Shenzhen, Guangdong
  - Sun Yat-sen University Cancer Center Internal medicine department, Guandong, Guangzhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Chenzhou first people's Hospital, Chenzhou, Hunan
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital Of Shandong University, Jinan, Shandong
  - Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality
  - The first Affiliated Hospital Of Xi'an Jiaotong University, Xi’an, Shanxi
  - The Second Affiliated Hospital Of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The first affiliated Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang